CLINICAL TRIAL: NCT06111352
Title: Outcome of OPC Poisoning Patients Between Two Treatment Groups One With Atropine Plus Pralidoxime and Other With Only Atropine
Brief Title: Outcome of Moderate Severity in OPC Poisoning Patients When Treated With Pralidoxime
Acronym: OPC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sir Salimullah Medical College Mitford Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Md. Mahmudul Hasan, MBBS, Medical officer, Sir salimullah Medical College Mitford Hospital, Dhaka, Bangladesh, Sir Salimullah Medical College Mitford Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 59.18.1100.031.18.011.22.2268
Record Dates: First submitted 2023-10-21; First posted 2023-11-01 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Organophosphorus Poisoning
MeSH Terms: conditions — Organophosphate Poisoning | interventions — pralidoxime; Atropine

STUDY DESIGN:
Intervention Model Description: Open level, Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Patients will be treated with Atropine plus pralidoxime
  Pralidoxime: Dosage:1gram; Dosage form: Intravenous infusion; Frequency: 8 hourly
  Atropine:
  Interventions: Drug: Pralidoxime; Drug: Atropine
- Group B (Other): Patients will be treated with only atropine
  Interventions: Drug: Atropine

INTERVENTIONS:
Drug: Pralidoxime — Inj. Pralidoxime 1 gm I/V will be given as first dose over 10-20 minutes. If no improvement of muscle weakness, then repeat the dose after one hour. Then 1 gram of Inj. Pralidoxime will be given at an 8-hour interval
  Arms: Group A
Drug: Atropine — Inj. Atropine (3 ampule) will be given in intravenous route as a first dose, rapidly. Then the dose will be doubled from the previous dose in every 5 minutes interval until the signs of atropinisation appeared. Then infusion of 10% of the total bolus dose (the dose that was given until the signs of atropinisation appeared) per hour, will be given with intravenous Normal saline/ 5% DNS(Dextrose and Sodium chloride) as a maintenance dose. The dose will be reduced for adjustment, based on clinical features/improvement

SUMMARY:
This open level randomized controlled trial will be conducted in the department of medicine at Sir Salimullah Medical College and Mitford Hospital. Clinical severity will be assessed by the POP (Peradeniya Organophosphorus Poisoning) scale of admitted patients having a history of organophosphorus poisoning within 24 hours with clinical features and physical evidence of poisoning consumed. Only moderate severity (POP Scale score 4-7) of OPC (Organophosphorus compound) patients will be included in this study. Then one group of patients will be treated with atropine and pralidoxime and another group will be treated with atropine. The outcome will be noted as clinical improvement or recovery. hospital stay, requirement of ICU, death.

DETAILED DESCRIPTION:
OPC poisoning is one of the most medical emergencies manage in hospital in our country. For the treatment of this acute cases, along with the supportive measures, intravenous anticholinergic atropine is the mostly used antidote. WHO (World Health Organization) recommended the use of intravenous pralidoxime along with atropine for favorable outcomes, while several studies had doubted effectiveness of its use for the treatment of OPC poisoning. Therefore, the aim of this study is assessment of the outcomes of patients with OPC poisoning of moderate severity between two treatment groups one will be treated with atropine plus Pralidoxime and other with only atropine. This open level randomized controlled trail will be conducted in department of Medicine, Sir Salimullah Medical College & Mitford Hospital, Dhaka. All the patient admitted in the hospital during the study period with OPC poisoning will be evaluated by clinical presentation. Form the total patients, those patients with the history of organophosphorus poisoning within previous 24 hours with clinical features of poison consumption with moderate severity after assessing by Peradeniya OP (POP) Scale and considering the inclusion and exclusion criteria; participant/patients will be enrolled in the study. A total 96 patients will be enrolled in the study. After inclusion in the study the participant will be randomly allocated following simple randomization technique in both treatment group [atropine plus pralidoxime group (Group A) and atropine only group (Group B). The nature of the chemical composition of the organophosphorus compound will be identified from the brought sample.

The patients of group (A) will be treated with atropine plus pralidoxime and all the patients of group (B) will be treated with atropine only. All patients will receive other supportive therapy with stomach wash, i.v. fluid, antibiotics, and O2 inhalation as required. Every patient will be followed up by careful clinical examination. Patients developing respiratory failure will be identified by clinical examination and by using pulse oximetry. These Patients will be treated in ICU of Sir Salimullah Medical College & Mitford Hospital and assisted ventilation support will be given. Both groups will be further analyzed from the start of poisoning to arrival at hospital and up to recovery/ ICU support/Death.

Each ampoule of inj atropine contained 0.6 mg atropine sulphate and each vial of inj. pralidoxime contained pralidoxime 1gm. Both drugs will be used in iv route. Inj. pralidoxime will be given as intravenous infusion over 4 minutes to avoid hypotension. Both antidotes will be administered as per recommended dosage schedule.

Inj. Atropine (3 ampule) will be given in intravenous route as a first dose, rapidly. Then the dose will be doubled from the previous dose in every 5 minutes interval until the signs of atropinisation appeared. Then infusion of 10% of the total bolus dose (the dose that was given until the signs of atropinisation appeared) per hour, will be given with intravenous Normal saline/ 5% DNS(Dextrose and Sodium chloride infusion) as a maintenance dose. The dose will be reduced for adjustment, based on clinical features/improvement. Inj. Pralidoxime 1 gm I/V will be given as first dose over 10-20 minutes. If no improvement of muscle weakness, then repeat the dose after one hour. Then 1 gram of Inj. Pralidoxime will be given at an 8-hour interval. The atropine and pralidoxime dose will be continued until symptomatic improvement and recovery. After discontinue of antidote further patient will be observed 24-48 hours then patient will be discharge. Study outcomes will provide any benefit of pralidoxime in moderately severe OPC poisoning patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient having history of organophosphorus poisoning within 24 hours with features of moderate severity. (POP scale score 4-7)
2. Age above 12 years

Exclusion Criteria:

1. Mixed poisons along with organophosphorus compound,
2. Patients with known case chronic diseases such as chronic lung disease, chronic kidney disease, Heart failure, malignancy, chronic liver disease

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Mortality rate | 1 year

SECONDARY OUTCOMES:
Proportion of patients who required intubation | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Salimullah Medical College Mitford Hospital, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No
I have some resource problem.